CLINICAL TRIAL: NCT03372772
Title: Effect of Levocarnitine Supplementation for the Management of Fatigue in Levothyroxine-Treated Hypothyroid Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh (Other)
Responsible Party: Principal Investigator, Dr. Farjana Akhter, Resident ( Phase-B), Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: No. BSMMU/2017/2668
Record Dates: First submitted 2017-12-10; First posted 2017-12-14 (Actual); Last update posted 2017-12-26 (Actual); Status verified 2017-12

CONDITIONS: Patient Compliance
Keywords: Fatigue, Levocarnitine,
MeSH Terms: conditions — Patient Compliance; Fatigue | interventions — Carnitine

STUDY DESIGN:
Intervention Model Description: Control Group- Patients with only levothyroxine therapy Interventional Group- Patients with Levocarnitine supplementation in addition to levothyroxine therapy
Who Masked: Participant
Masking Description: Single Blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (No Intervention): Control group - patients with only levothyroxine therapy
- Intervention group (Experimental): Intervention Group- Patients with levocarnitine supplementation in addition to levothyroxine therapy
  Interventions: Drug: Levocarnitine

INTERVENTIONS:
Drug: Levocarnitine — Levocarnitine syrup- Oral supplementation about 2000mg/ day for 8 weeks
  Other Names: Levocarnitine syrup
  Arms: Intervention group

SUMMARY:
It has been observed that despite administration of apparently adequate thyroid hormone replacement in hypothyroid patients, many of them experience persistent fatigue and fatigue-related symptoms. Carnitine transports long chain fatty acids into the mitochondria whereupon the high energy source (ATP) becomes synthesized. Levocarnitine administration reduced fatigue related symptoms in hypothyroid patients receiving thyroid hormone replacement. The present study deals with alleviation of fatigue in hypothyroid patients by carnitine supplementation.

DETAILED DESCRIPTION:
It has been well-established now-a-days that, some chronic diseases impose generalized weakness, lethargy, lassitude amounting from degrees mild, moderate to a severe one to total incapacitation on the part of the patients. Hypothyroid patients instate of receiving adequate thyroid hormone replacement, experience fatigue-related symptoms. Carnitine is a non-essential amino acid synthesized endogenously from essential amino acids- lysine and methionine with in the body involved in long chain fatty acid transportation to the mitochondrial membrane. Carnitine- transportation system is essential for production of energy at cellular level. Thyroid hormone plays an important role in carnitine-dependent long chain fatty acid transport and oxidation. Some available reports suggest that, Levocarnitine supplementation produced potentially favourable effects on fatigue-related symptoms in hypothyroid patients although still awaits confirmation. The present study is an attempt to investigate into the effects of Levocarnitine supplementation on fatigue in patients with hypothyroidism.

ELIGIBILITY:
Inclusion Criteria:

i. Clinical diagnosis of primary hypothyroidism patients with fatigue symptoms ii. Age : From 20 to 50 years iii. Levothyroxine treatment: receiving for at least 6 months iv. Serum free thyroxine level: 0.80-1.80 ng/dl v. Serum Thyroid-stimulating hormone level: 0.35-5.50 µIU/ml ( µIU = micro international unit)

-

Exclusion Criteria:

i. Patients with Hypothyroidism 20 years and 50 years ii. Acute or chronic liver diseases iii. Anaemia iv. Clinical diagnosis of Diabetes mellitus. v. Cardiovascular disease ( such as heart failure, arrhythmia and uncontrolled hypertension ) vi. Patients with psychological disorders (such as depression, anxiety disorder, schizophrenia, alcoholism or fatigue disorder due to other systemic diseases) vii. Patients having serious infections or terminal illness (such as tuberculosis, HIV or malignant tumor ) viii. Autoimmune diseases ( such as rheumatoid arthritis, Systemic lupus erythematosus or multiple sclerosis) ix. Patients with impaired renal function x. Pregnant or planned to be pregnant xi. Nursing mothers

-

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2017-03-16 (Actual); Primary Completion 2017-12-30 (Estimated); Study Completion 2018-02-28 (Estimated)

PRIMARY OUTCOMES:
Fatigue score | 8 weeks
  Alleviation of fatigue level

SECONDARY OUTCOMES:
Lipid profile | 8 weeks
  Effect of Levocarnitine on lipid level

CONTACTS AND LOCATIONS:
Overall Officials: Farjana Akhter, MBBS, Principal Investigator — Resident ,Phase-B
Locations (1):
- Phamacology Department, BSMMU, Dhaka, Shahbag, Bangladesh

IPD SHARING:
Plan to Share IPD: No